CLINICAL TRIAL: NCT01747200
Title: Modulating Behavior in Humans by Entrainment With Rhythmic Transcranial Magnetic Stimulation
Brief Title: Effects of Transcranial Magnetic Stimulation on Object Recognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Purpose: Basic Science
Other Study IDs: 130035; 13-N-0035
Record Dates: First submitted 2012-12-08; First posted 2012-12-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-01-26

CONDITIONS: Repetitive TMS (rTMS); Sham rTMS; Bilateral rTMS; Unilateral rTMS
Keywords: Repetitive TMS (rTMS)

INTERVENTIONS:
Procedure: Sham rTMS
Procedure: Bilateral rTMS at same frequency and in phase
Procedure: Bilateral rTMS at different frequencies
Procedure: Bilateral rTMSat same frequency and out of phase
Procedure: rTMS over TP8
Procedure: rTMS over TP7

SUMMARY:
Background:

- The brain has natural rhythms called brain waves. An electroencephalogram (EEG) can record these rhythms. When people identify the picture of a familiar object shown on a computer screen, the communication between certain regions of the brain increases. An EEG can detect these communication brain waves. Transcranial magnetic stimulation (TMS) can affect these brain waves by slightly changing the brain s rhythms. Researchers want to see if changing brain rhythms with TMS interferes with the ability to identify pictures of familiar objects. This study will provide more information about how TMS can affect brain waves and behavior.

Objectives:

- To see if TMS can interfere with the brain s ability to identify pictures of familiar objects.

Eligibility:

- Healthy volunteers between 18 and 70 years of age.

Design:

* This study requires two visits to the clinical center. The first visit will last about 2 hours. The second visit will last about 4 hours.
* Participants will be screened with a physical exam and medical history.
* At the first visit, participants will have an object recognition test. Participants will look at pictures of several objects on a computer screen. They will then have to state whether the objects they see on the screen are familiar. The object recognition test will be done along with TMS.
* At the second visit, participants will have an EEG while taking the object recognition test. Brain waves will be monitored during the test. They will then repeat the test while having repetitive TMS to study its effect on object recognition. The participants will then take the object recognition test alone for a final time. This will make sure that TMS effects (if any) on the ability to identify familiar object images are no longer present.

DETAILED DESCRIPTION:
Inter-hemispheric coherence (IHC) is one of the electroencephalography (EEG) parameters that measures synchronization of oscillations originating from brain regions of different hemispheres and thereby the functional connectivity between them. We know that object discrimination is associated with transient increase in IHC. In this study we will interfere with the transient IHC that is associated with midline object discrimination by using rhythmic repetitive transcranial magnetic stimulation (rTMS).

We will study the effects of entrainment by unilateral or bilateral, synchronous or asynchronous TMS pulses on behavior. The goal of the study is to determine if entrainment by TMS will affect task performance. If the results show that TMS by entrainment influenced behavior, then we can expect TMS to be a useful technique to explore the behavioral impact of specific neuronal oscillations under physiological as well as pathological conditions. Further, TMS could also find applications in rehabilitation or treatment of behavioral symptoms in patients with neuropsychiatric diseases.

STUDY POPULATION:

We intend to study 11 adult healthy volunteers on an outpatient basis.

STUDY DESIGN:

All the subjects will first participate in a screening session where the threshold TMS intensity for blocking object discrimination and the optimal coil orientation will be determined using single pulse TMS. Later they will attend the main experiment session where they will be asked to perform the object discrimination task in four blocks, of which the second, third and fourth will be in random order. During the first block, the individual coherence frequency will be determined by recording EEG during the task. During the second, third and fourth blocks, the subjects will receive either unilateral, bilateral or sham rTMS in a random order while EEG is being recorded. Short trains of 7 TMS pulses will be delivered during each trial. TMS pulses will be administered over left and/or right LOG at 80% of threshold intensity blocking object discrimination or 60% maximum stimulator output whichever is smaller.

OUTCOME MEASURES:

We expect that short trains of TMS will affect IHC depending on whether the pulses are synchronous or asynchronous. By modulating IHC, we expect changes in object discrimination task performance. The primary outcome measure in this study includes object discrimination task performance. During the study, we will also compute the individual frequency at which maximum coherence occurs, the threshold intensity and optimal coil direction for blocking object discrimination and the spatio-temporal characteristics of EEG waves during the rTMS trains to confirm that entrainment is occurring.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age between 18 - 70 years.
* Able to give his/her own consent to participate in the study.

EXCLUSION CRITERIA:

* Presence of cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain, cochlear implants, metal fragments in the eye.
* Pregnancy or lactation.
* History of any serious medical illness or hearing problems
* Intake of medication that affect the central nervous system like anti depressants, antihistamines, antipsychotics, dopamine agonists, benzodiazepines and antiepileptics in the past 3 months.
* Presence of neurological or psychiatric illnesses like brain tumor, migraine, depression, bipolar disorder, schizophrenia.
* History of any seizure.
* Use or abuse of any drug in the past 6 months or intake of more than 7 alcoholic drinks a week in females and more than 14 alcoholic drinks a week in males.

Exclusion criteria specific for MRI::

* Presence of metal in the body, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain or on blood vessels, cochlear implants, artificial heart valves or metal fragments in the eye as these make having an MRI unsafe.
* Presence of metallic dental fillings which are likely to cause MRI artifacts
* Uncomfortable being in a small space for up to 2 hours.
* Unable to lie flat on the back for up to 2 hours

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-11-16; Primary Completion 2017-01-26 (Actual); Study Completion 2017-01-26 (Actual)

PRIMARY OUTCOMES:
Percentage of correct responses in the midline object recognition task. | 4 hours

SECONDARY OUTCOMES:
Threshold intensity for blocking object recognition | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adler G, Brassen S, Jajcevic A. EEG coherence in Alzheimer's dementia. J Neural Transm (Vienna). 2003 Sep;110(9):1051-8. doi: 10.1007/s00702-003-0024-8. PMID 12928837
- [Background] Gerloff C, Andres FG. Bimanual coordination and interhemispheric interaction. Acta Psychol (Amst). 2002 Jun;110(2-3):161-86. doi: 10.1016/s0001-6918(02)00032-x. PMID 12102104
- [Background] Gray CM, Singer W. Stimulus-specific neuronal oscillations in orientation columns of cat visual cortex. Proc Natl Acad Sci U S A. 1989 Mar;86(5):1698-702. doi: 10.1073/pnas.86.5.1698. PMID 2922407